CLINICAL TRIAL: NCT03068234
Title: A Randomized, Double-blinded, Placebo Controlled Study to Evaluate Clinical Efficacy and Safety of Pirfenidone for Skin Fibrosis in Systemic Sclerosis
Brief Title: Pirfenidone as Treatment of Skin Fibrosis in Systemic Sclerosis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: [2017]17
Record Dates: First submitted 2017-02-16; First posted 2017-03-01 (Actual); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic | interventions — pirfenidone; Steroids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pirfenidone group (Experimental): The subjects will receive pirfenidone from 200mg three times a day, oral administrated, with low dose steroids.
  Interventions: Drug: Pirfenidone; Drug: Steroids
- Control group (Placebo Comparator): The subjects will receive placebo within first 24-week, and pirfenidone 200mg three times a day for the second 24-week, with low dose steroids.
  Interventions: Drug: Pirfenidone; Drug: Placebo oral capsule; Drug: Steroids

INTERVENTIONS:
Drug: Pirfenidone — A chemical synthesized agent showing anti-fibrotic effects in idiopathic pulmonary fibrosis.
Drug: Placebo oral capsule — Placebo for pirfenidone capsule
  Arms: Control group
Drug: Steroids — Low dose of glucocorticoids, a basic treatment for patients with systemic sclerosis

SUMMARY:
This study is to evaluate the efficacy and safety of an antifibrotic agent, pirfenidone as treatment of systemic sclerosis. The primary outcome of this study is improvement of skin fibrosis.

DETAILED DESCRIPTION:
All patients enrolled should suffer from moderate to severe skin fibrosis at the screening stage.

The study period is 52 week. The study contains two stages, a 24-week blind stage following with open stage for another 24-week period of time. Subjects will receive pirfenidone or placebo randomized in the first 24-week and will all receive pirfenidone treatment in the second 24-week, with of combination of low dose steroids.

The secondary outcomes of this study include but not limit to safety, improvement of lung fibrosis and digital ulcer burden.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill EULAR/ACR classification criteria (2013) for systemic sclerosis (SSc).
* Subjects must have mRSS≥10 at screening stage
* Subjects must have signs of fibrosis in their chest CT at screening stage
* If a subject has received treatments before, it should be stable at least 3 months until screening and with no significant efficacy (ΔmRSS≤-2)

Exclusion Criteria:

* Subjects with other connective tissue diseases overlapping with SSc
* Subjects with skin atrophy as the main cutaneous manifestation
* Subjects with active digital ulcers or gangrene
* Active severe SSc-driven renal disease or heart dysfunction at screening
* Subjects with significant hematologic abnormalities
* Abnormal liver function test at screening (ALT, AST or total bilirubin over 2 fold of upper normal level
* Clinically significant active infection including ongoing and chronic infections
* History of human immunodeficiency virus (HIV)
* Confirmed Positive tests for hepatitis B or positive test for hepatitis C
* Active tuberculosis
* Live or attenuated vaccine within 4 weeks prior to screening
* Subjects with significant hematologic abnormalities

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Modified Rodnan Skin Score (mRSS） | Week 52
  A semi-quantitative score for skin fibrosis of every subjects

SECONDARY OUTCOMES:
Modified Rodnan Skin Score | Week 24
  A semi-quantitative score for skin fibrosis of every subjects
Assessment of chest CT | Week 52
  Semi-quantitative scale for fibrotic changes in chest CT images from an individual patient
Assessment of chest CT | Week 24
  Semi-quantitative scale for fibrotic changes in chest CT images from an individual patient
Forced vital capacity | Week 52
  A marker for lung function that may decrease with pulmonary fibrosis
Forced vital capacity | Week 24
  A marker for lung function that may decrease with pulmonary fibrosis
Diffusing capacity | Week 52
  Another marker for lung function that may decrease with pulmonary fibrosis
Diffusing capacity | Week 24
  Another marker for lung function that may decrease with pulmonary fibrosis
6 minute walk test | Week 52
  A simple, well-accepted and quantitative clinical exam to test heart and lung function
6 minute walk test | Week 24
  A simple, well-accepted and quantitative clinical exam to test heart and lung function
Hand function assessment | Week 52
  Hand function will be measured by Cochin Hand Function Scale
Hand function assessment | Week 24
  Hand function will be measured by Cochin Hand Function Scale
Proportion of subjects with increased mRSS | Week 52
  Proportion of subjects with ∆mRSS≥5
Proportion of subjects with increased mRSS | Week 24
  Proportion of subjects with ∆mRSS≥5
Quality of life | Week 52
  Assessed by the health assessment questionnaire disability index
Quality of life | Week 24
  Assessed by the health assessment questionnaire disability index
Safety and Tolerability | Week 52
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Safety and Tolerability | Week 24
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- RenJi Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided